CLINICAL TRIAL: NCT05775692
Title: Beijing Chilrens' Hospital
Brief Title: Population Pharmacokinetics of Fluconazole in the Treatment of Neonatal Fungal Infectious Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Adong Shen, Deputy Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: NCT2020
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Fluconazole; Infection; Newborn; Pharmacokinetics
MeSH Terms: conditions — Infections | interventions — Fluconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — whole blood and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns and children with the usage of fluconazole: Newborn with fluconazole against infectious diseases.
  Interventions: Drug: fluconazole

INTERVENTIONS:
Drug: fluconazole — According to the models of population pharmacokinetics,the investigators and want to correlate use of fluconazole with treatment effectiveness and safety in newborns

SUMMARY:
This study is based on the hypothesis that the pharmacokinetics of fluconazole in newborns and children are different from adults. We aim to study the population pharmacokinetics of newborns and children receiving the fluconazole for treatment of infectious diseases. In this study, we will detect fluconazole concentration in plasma by using residual blood samples of blood gas analysis and other clinical tests and employ computers for constructing population pharmacokinetic models. In addition, we also want to correlate use of fluconazole with treatment effectiveness and incidence of adverse effects in newborns and children. This novel knowledge will allow better and more rational approaches to the treatment of infectious diseases in newborns and children. It will also set the foundation for further studies to improve fluconazole therapies for newborns and children.

DETAILED DESCRIPTION:
1. Establish population pharmacokinetic (PPK) models of fluconazole in newborns and children by nonlinear mixed effect modeling (NONMEM).

   At different timepoint after fluconazole administration, plasma samples of 50 newborns and children will be collected from neonatal intensive care unit (NICU) and pneumology department for fluconazole. The clinical information includes demography, medication, concentration data, blood biochemical parameters and so on .

   Plasma samples will be tested by high performance liquid chromatography (HPLC). PPK models of fluconazole will be established by NONMEM program. The reliability and stability of the PPK model will be evaluated by 1000 times of Bootstrap procedure and normalized predictive distribution error (NPDE).
2. Evaluation of the clinical feasibility and safety of individualized dosing.

According the results of PPK models, we will use dosages recommended in models to cure children infectious diseases in prospective studies. For fluconazole, 150 newborns and children will be collected.

We will compare the therapeutic effects and safety between newborns and children with conventional therapies and those with individualized therapies, including proportions of newborns and children with effective fluconazole concentration, improvement speed of of newborns and children, liver and kidney functions, adverse reactions of drugs, and so on.

ELIGIBILITY:
Inclusion Criteria:

Newborn （0-28d） with fluconazole against infectious diseases. The anti-infective therapy includes drugs commonly used in children infectious diseases.

Newborns infectious diseases include pneumonia, sepsis, purulent meningitis and other diseases with infection.

Informed consent signed by the parents and/or guardians.

Exclusion Criteria:

1. Allergic to any class of antibiotics;
2. Receiving other experimental drugs;
3. There are other factors that clinicians consider unsuitable for inclusion in the study.

Ages: 1 Minute to 28 Days | Sex: All
Age Groups: Child
Gender Based: Yes
Study Population: Neonates on fluconazole
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | up to 4 weeks
  Cmax is a term used in pharmacokinetics refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose.

CONTACTS AND LOCATIONS:
Overall Officials: A-Dong Shen, Master, Principal Investigator — Beijing Children's Hospital of Capital Medical University
Locations (1):
- Beijing Children's Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao W, Lopez E, Biran V, Durrmeyer X, Fakhoury M, Jacqz-Aigrain E. Vancomycin continuous infusion in neonates: dosing optimisation and therapeutic drug monitoring. Arch Dis Child. 2013 Jun;98(6):449-53. doi: 10.1136/archdischild-2012-302765. Epub 2012 Dec 19. PMID 23254142
- [Background] Leroux S, Zhao W, Betremieux P, Pladys P, Saliba E, Jacqz-Aigrain E; French Society of Neonatology. Therapeutic guidelines for prescribing antibiotics in neonates should be evidence-based: a French national survey. Arch Dis Child. 2015 Apr;100(4):394-8. doi: 10.1136/archdischild-2014-306873. Epub 2015 Jan 27. PMID 25628457
- [Background] Jacqz-Aigrain E, Leroux S, Zhao W, van den Anker JN, Sharland M. How to use vancomycin optimally in neonates: remaining questions. Expert Rev Clin Pharmacol. 2015;8(5):635-48. doi: 10.1586/17512433.2015.1060124. Epub 2015 Aug 4. PMID 26289222